CLINICAL TRIAL: NCT03360149
Title: Health Practice of Hemophilia Patiente Care During Pregnancy, Delivery and Newborn Children
Acronym: ECHANGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ECHANGE
Record Dates: First submitted 2017-10-19; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Hemophilia
Keywords: Hemophilia pregnant; Hemophilia delivery; Hemophilia children
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prenancy and specialy delivery for hemophilia mother and her children possibly hemophilia is risked.

Diagnostical of hemophilia pregnan is the first difficulty but patients with hemorrhagic menstruation without etiology known, hemorrhagic complication during a chirurgical procedure or during previously pregnancy currently are examine in Haemostasis consultation.

None French recommendation specifie for health practice of these hemophilia patients exists. However, Anglo-Saxon recommendations are published in 2011.

The objective of this study is to realize a French investigation of health practice about hemophilia care of these patients and to compare them with the English reference table.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Hemophilia A or B
* Pregnancy between 2014 and 2016

Exclusion Criteria:

- Opposition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult with Hemophilia A or B during Pregnancy, Delivery and Newborn Children
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
antenatal care in pregnant women carriers of hemophilia | during pregnancy
  Frequency of Diagnosis
labour and delivery procedures | day of delivery
  childbirth procedure type
post-partum care | day of delivery until 3 month
  treatment type
children care | day of delivery until 3 month
  complication type
antenatal care in pregnant women carriers of hemophilia | 9 month (during pregnancy)
  description of complications
antenatal care in pregnant women carriers of hemophilia | 9 month (during pregnancy)
  patient follow up
labour and delivery procedures | day of delivery
  therapeutic protocol type
labour and delivery procedures | day of delivery
  analgesic type
labour and delivery procedures | day of delivery
  blood loss measurement
post-partum care | day of delivery until 3 month
  feeding
post-partum care | day of delivery until 3 month
  contraception type
post-partum care | day of delivery until 3 month
  time of menses returns
children care | day of delivery until 3 month
  hemophilia diagnostic
children care | day of delivery until 3 month
  treatment type

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU d'Angers, Angers
  - CHRU de Brest, Brest
  - Ch Le Mans, Le Mans
  - CHU de Nantes, Nantes
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU de TOURS, Tours

REFERENCES:
- [Derived] Nau A, Gillet B, Guillet B, Beurrier P, Ardillon L, Cussac V, Guillou S, Raj L, Trossaert M, Horvais V, Bayart S, Potin J, Rose J, Macchi L, Couturaud F, Lacut K, Pan-Petesch B. Bleeding complications during pregnancy and delivery in haemophilia carriers and their neonates in Western France: An observational study. Haemophilia. 2020 Nov;26(6):1046-1055. doi: 10.1111/hae.14117. Epub 2020 Aug 25. PMID 32842170